CLINICAL TRIAL: NCT01094366
Title: An Evaluation of the Paracervical Block for Pain Control in First Trimester Surgical Abortion
Brief Title: Paracervical Block for Pain Control in First Trimester Abortion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Planned Parenthood Federation of America (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: OHSU IRB 6071
Record Dates: First submitted 2010-03-25; First posted 2010-03-26 (Estimated); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Legal Abortion With Complication; Pain
Keywords: Paracervical Block; pain control; abortion
MeSH Terms: conditions — Pain; Agnosia | interventions — Anesthesia, Obstetrical

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Paracervical Block for Pain Control (Sham Comparator): Subject will not receive a paracervical block during the procedure
  Interventions: Procedure: Sham Paracervical Block
- Paracervical Block for Pain Control (Active Comparator): Subject will receive a paracervical block during the procedure.
  Interventions: Procedure: Paracervical Block

INTERVENTIONS:
Procedure: Paracervical Block — Subject receives 20 mL paracervical block with 18 mL of 1% Lidocaine solution buffered with 2 mL 8.4% sodium bicarbonate for pain control.
  Arms: Paracervical Block for Pain Control
Procedure: Sham Paracervical Block — In the non-intervention group, the surgeon performs a sham PCB during which 2 mL buffered lidocaine solution are injected at the tenaculum site, after which a capped needle gently simulates the standard PCB procedure.
  Arms: No Paracervical Block for Pain Control

SUMMARY:
Many woman undergoing a surgical abortion receive a paracervical nerve block for pain reduction, in which lidocaine (a numbing medication) is injected around the cervix. These injections numb the cervix and possibly the lower part of the uterus. However, the injection can be uncomfortable and it is not well known whether it is effective in reducing pain. The purpose of this study is to determine the level of pain women experience with a surgical abortion and the effect that paracervical block might have on that pain.

DETAILED DESCRIPTION:
The investigators expect to have 120 women complete this study, between study sites at OHSU's Center for Women's Health and Planned Parenthood Columbia Willamette in Portland, OR. Every participant will still receive the standard oral medication for pain (ibuprofen) and anxiety (lorazepam). Eligible subjects will be at least 18 years of age, less than 11 weeks pregnant and have already decided to have a surgical abortion.

The primary outcome evaluated will be pain reported at time of cervical dilation. The investigators will assess pain at various time points (including secondary outcomes) immediately upon completion of the respective step and pain and satisfaction 30 minutes postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or older
* Voluntarily requesting pregnancy termination
* Ultrasound confirmed intrauterine pregnancy up to 10 6/7 weeks gestational age
* Good general health
* English or Spanish speaking
* Be able and willing to sign an informed consent and agree to terms of the study

Exclusion Criteria:

* Gestational ages over 11 0/7 weeks, due to routine misoprostol use at our institutions
* Incomplete abortion
* Required or requested narcotics or IV sedation (prior to randomization)
* Patients who refuse Ibuprofen and paracervical blocks
* Contraindications or allergies to lidocaine, ibuprofen or ativan
* Significant physical or mental health condition
* Adnexal mass or tenderness on pelvic exam consistent with pelvic inflammatory disease
* Patients with known hepatic disease
* Women, who in the opinion of the investigator are not suitable for the study protocol

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2010-04; Primary Completion 2010-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Pain reported with cervical dilation | 1 Year
  Distance (mm) from the left of the 100-mm VAS scale (reflecting magnitude of pain) recorded at time of cervical dilation.

SECONDARY OUTCOMES:
Anticipated and reported pain at various time points | 1 Year
  Distance (mm) from the left of the 100-mm VAS scale (reflecting magnitude of anticipated pain) recorded prior to the procedure.
  Distance (mm) from the left of the 100-mm VAS scale (reflecting magnitude of pain) recorded at time of positioning for procedure, speculum insertion, placement of the PCB, aspiration and 30 min postoperatively.
Anxiety reported with the pain expected during the procedure and the procedure itself. | 1 Year
  Distance (mm) from the left of the 100-mm VAS scale (reflecting degree of anxiety) recorded prior to procedure.
Satisfaction reported with pain control and overall procedure | 1 Year
  Distance (mm) from the left of the 100-mm VAS scale (reflecting degree of satisfaction) recorded post procedure.
Need for additional intraoperative and/or postoperative pain medication | 1 Year
  Subjects may request additional pain medication once their procedure has begun or in recovery. The need for additional medication, and what medication was subsequently distributed, will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Regina M Renner, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Planned Parenthood Columbia Willamette, Portland, Oregon, United States

REFERENCES:
- [Background] Allen RH, Kumar D, Fitzmaurice G, Lifford KL, Goldberg AB. Pain management of first-trimester surgical abortion: effects of selection of local anesthesia with and without lorazepam or intravenous sedation. Contraception. 2006 Nov;74(5):407-13. doi: 10.1016/j.contraception.2006.06.002. Epub 2006 Aug 2. PMID 17046383
- [Background] Belanger E, Melzack R, Lauzon P. Pain of first-trimester abortion: a study of psychosocial and medical predictors. Pain. 1989 Mar;36(3):339-350. doi: 10.1016/0304-3959(89)90094-8. PMID 2710563
- [Background] Berger GS, Tyler CW, Harrod EK. Maternal deaths associated with paracervical block anesthesia. Am J Obstet Gynecol. 1974 Apr 15;118(8):1142-3. doi: 10.1016/0002-9378(74)90698-x. No abstract available. PMID 4817653
- [Background] Blanco LJ, Reid PR, King TM. Plasma lidocaine levels following paracervical infiltration for aspiration abortion. Obstet Gynecol. 1982 Oct;60(4):506-8. PMID 7121936
- [Background] Cetin A, Cetin M. Effect of deep injections of local anesthetics and basal dilatation of cervix in management of pain during legal abortions. A randomized, controlled study. Contraception. 1997 Aug;56(2):85-7. doi: 10.1016/s0010-7824(97)00096-6. PMID 9315416
- [Background] Donati S, Medda E, Proietti S, Rizzo L, Spinelli A, Subrizi D, Grandolfo ME. Reducing pain of first trimester abortion under local anaesthesia. Eur J Obstet Gynecol Reprod Biol. 1996 Dec 27;70(2):145-9. doi: 10.1016/s0301-2115(95)02583-9. PMID 9119094
- [Background] Edelman A, Nichols MD, Leclair C, Astley S, Shy K, Jensen JT. Intrauterine lidocaine infusion for pain management in first-trimester abortions. Obstet Gynecol. 2004 Jun;103(6):1267-72. doi: 10.1097/01.AOG.0000127981.53911.0e. PMID 15172863
- [Background] Edelman A, Nichols MD, Leclair C, Jensen JT. Four percent intrauterine lidocaine infusion for pain management in first-trimester abortions. Obstet Gynecol. 2006 Feb;107(2 Pt 1):269-75. doi: 10.1097/01.AOG.0000194204.71925.4a. PMID 16449111
- [Background] Glantz JC, Shomento S. Comparison of paracervical block techniques during first trimester pregnancy termination. Int J Gynaecol Obstet. 2001 Feb;72(2):171-8. doi: 10.1016/s0020-7292(00)00292-7. PMID 11166751
- [Background] Gomez PI, Gaitan H, Nova C, Paradas A. Paracervical block in incomplete abortion using manual vacuum aspiration: randomized clinical trial. Obstet Gynecol. 2004 May;103(5 Pt 1):943-51. doi: 10.1097/01.AOG.0000123269.86525.c4. PMID 15121569
- [Background] Grimes DA, Cates W Jr. Deaths from paracervical anesthesia used for first-trimester abortion, 1972-1975. N Engl J Med. 1976 Dec 16;295(25):1397-9. doi: 10.1056/NEJM197612162952503. PMID 980095
- [Background] Hakim-Elahi E, Tovell HM, Burnhill MS. Complications of first-trimester abortion: a report of 170,000 cases. Obstet Gynecol. 1990 Jul;76(1):129-35. PMID 2359559
- [Background] Jensen MP, Chen C, Brugger AM. Interpretation of visual analog scale ratings and change scores: a reanalysis of two clinical trials of postoperative pain. J Pain. 2003 Sep;4(7):407-14. doi: 10.1016/s1526-5900(03)00716-8. PMID 14622683
- [Background] Kan AS, Caves N, Wong SY, Ng EH, Ho PC. A double-blind, randomized controlled trial on the use of a 50:50 mixture of nitrous oxide/oxygen in pain relief during suction evacuation for the first trimester pregnancy termination. Hum Reprod. 2006 Oct;21(10):2606-11. doi: 10.1093/humrep/del234. Epub 2006 Jun 21. PMID 16790607
- [Background] Kan AS, Ng EH, Ho PC. The role and comparison of two techniques of paracervical block for pain relief during suction evacuation for first-trimester pregnancy termination. Contraception. 2004 Aug;70(2):159-63. doi: 10.1016/j.contraception.2004.03.013. PMID 15288222
- [Background] Lopez JC, Vigil-De Gracia P, Vega-Malek JC, Ruiz E, Vergara V. A randomized comparison of different methods of analgesia in abortion using manual vacuum aspiration. Int J Gynaecol Obstet. 2007 Nov;99(2):91-4. doi: 10.1016/j.ijgo.2007.05.023. Epub 2007 Jul 12. PMID 17628562
- [Background] Miller L, Jensen MP, Stenchever MA. A double-blind randomized comparison of lidocaine and saline for cervical anesthesia. Obstet Gynecol. 1996 Apr;87(4):600-4. doi: 10.1016/0029-7844(95)00463-7. PMID 8602315
- [Background] Nichols, M. D., Halvorson-Boyd, G., Goldstein, R., Gevirtz, C., & Healow, D. (2009). Pain management. In M. Paul, E. S. Lichtenberg, L. Borgatta, D. A. Grimes & P. G. Stubblefield (Eds.), Management of unintended and abnormal pregnancy. (pp. 90-110): Wiley-Blackwell.
- [Background] O'Connell K, Jones HE, Simon M, Saporta V, Paul M, Lichtenberg ES; National Abortion Federation Members. First-trimester surgical abortion practices: a survey of National Abortion Federation members. Contraception. 2009 May;79(5):385-92. doi: 10.1016/j.contraception.2008.11.005. Epub 2008 Dec 11. PMID 19341852
- [Background] Owolabi OT, Moodley J. A randomized trial of pain relief in termination of pregnancy in South Africa. Trop Doct. 2005 Jul;35(3):136-9. doi: 10.1258/0049475054620923. PMID 16105333
- [Background] Phair N, Jensen JT, Nichols MD. Paracervical block and elective abortion: the effect on pain of waiting between injection and procedure. Am J Obstet Gynecol. 2002 Jun;186(6):1304-7. doi: 10.1067/mob.2002.123734. PMID 12066113
- [Background] Rabin JM, Spitzer M, Dwyer AT, Kaiser IH. Topical anesthesia for gynecologic procedures. Obstet Gynecol. 1989 Jun;73(6):1040-4. doi: 10.1097/00006250-198906000-00027. PMID 2657523
- [Background] Renner RM, Jensen JT, Nichols MD, Edelman A. Pain control in first trimester surgical abortion. Cochrane Database Syst Rev. 2009 Apr 15;2009(2):CD006712. doi: 10.1002/14651858.CD006712.pub2. PMID 19370649
- [Background] Rowbotham MC. What is a "clinically meaningful" reduction in pain? Pain. 2001 Nov;94(2):131-132. doi: 10.1016/S0304-3959(01)00371-2. No abstract available. PMID 11690725
- [Background] Smith GM, Stubblefield PG, Chirchirillo L, McCarthy MJ. Pain of first-trimester abortion: its quantification and relations with other variables. Am J Obstet Gynecol. 1979 Mar 1;133(5):489-98. doi: 10.1016/0002-9378(79)90282-5. PMID 443287
- [Background] Strauss LT, Gamble SB, Parker WY, Cook DA, Zane SB, Hamdan S; Centers for Disease Control and Prevention (CDC). Abortion surveillance--United States, 2004. MMWR Surveill Summ. 2007 Nov 23;56(9):1-33. PMID 18030283
- [Background] Suprapto K, Reed S. Naproxen sodium for pain relief in first-trimester abortion. Am J Obstet Gynecol. 1984 Dec 15;150(8):1000-1. doi: 10.1016/0002-9378(84)90399-5. PMID 6507524
- [Background] Todd KH, Funk KG, Funk JP, Bonacci R. Clinical significance of reported changes in pain severity. Ann Emerg Med. 1996 Apr;27(4):485-9. doi: 10.1016/s0196-0644(96)70238-x. PMID 8604867
- [Background] Safe Abortion: Technical and Policy Guidance for Health Systems. 2nd edition. Geneva: World Health Organization; 2012. Available from http://www.ncbi.nlm.nih.gov/books/NBK138196/ PMID 23700650
- [Background] Wiebe E, Podhradsky L, Dijak V. The effect of lorazepam on pain and anxiety in abortion. Contraception. 2003 Mar;67(3):219-21. doi: 10.1016/s0010-7824(02)00516-4. PMID 12618257
- [Background] Wiebe ER. Comparison of the efficacy of different local anesthetics and techniques of local anesthesia in therapeutic abortions. Am J Obstet Gynecol. 1992 Jul;167(1):131-4. doi: 10.1016/s0002-9378(11)91645-7. PMID 1442914
- [Background] Wiebe ER, Rawling M. Pain control in abortion. Int J Gynaecol Obstet. 1995 Jul;50(1):41-6. doi: 10.1016/0020-7292(95)02416-a. PMID 7556858
- [Background] Zullo F, Pellicano M, Stigliano CM, Di Carlo C, Fabrizio A, Nappi C. Topical anesthesia for office hysteroscopy. A prospective, randomized study comparing two modalities. J Reprod Med. 1999 Oct;44(10):865-9. PMID 10554747
- [Derived] Renner RM, Nichols MD, Jensen JT, Li H, Edelman AB. Paracervical block for pain control in first-trimester surgical abortion: a randomized controlled trial. Obstet Gynecol. 2012 May;119(5):1030-7. doi: 10.1097/AOG.0b013e318250b13e. PMID 22525915